CLINICAL TRIAL: NCT03446222
Title: Epicardial Mini-Maze Versus Catheter Ablation for the Management of Persistent Atrial Fibrillation
Acronym: EMMCAF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-15-0880
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catheter Ablation (Active Comparator): Catheter based radiofrequency ablation with wide antral circumferential PVI and isolation of posterior wall will be performed. Mitral and cavo-tricuspid isthmus ablation will be done only if such isthumus dependent flutters are documented prior to / during the procedure.
  Interventions: Procedure: Catheter ablation
- Mini-maze surgical procedure (Active Comparator): Wolf Mini-maze surgical ablation along with left atrial appendage ligation will be performed.
  Interventions: Procedure: Mini-maze surgical procedure

INTERVENTIONS:
Procedure: Catheter ablation — Catheter based radiofrequency ablation with wide antral circumferential PVI and isolation of posterior wall will be performed. Mitral and cavo-tricuspid isthmus ablation will be done only if such isthumus dependent flutters are documented prior to / during the procedure.
  Arms: Catheter Ablation
Procedure: Mini-maze surgical procedure — Wolf Mini-maze surgical ablation along with left atrial appendage ligation will be performed.
  Arms: Mini-maze surgical procedure

SUMMARY:
This study will assess the efficacy of catheter ablation versus the Wolf Mini-Maze surgical ablation for rhythm control in patients with persistent afib.

DETAILED DESCRIPTION:
Higher success rates have been achieved after a single surgical ablation when compared to catheter ablation, however contiguous and transmural lesions are not always guaranteed.

Even though, catheter ablation is now being offered for symptomatic persistent AF, recurrence after the index procedure in such a persistent AF substrate is not unusual. Redo-catheter ablation is routinely offered for such patients; however long term success still remains low. Non-pulmonary vein triggers are often targeted in such redo-catheter ablation procedures; though this approach remains controversial. More recently, the Wolf Mini-Maze procedure has been utilized with promising results.

This study proposes to randomize a group of persistent AF patients to undergo either catheter ablation or the surgical mini-maze procedure with left atrial appendage (LAA) ligation

ELIGIBILITY:
Inclusion Criteria:

* Persistent symptomatic AF with failure of at least 1 anti-arrhythmic drug
* Prior pulmonary vein isolation (PVI)
* CHA2DS2VASC > 0
* Able to tolerate and compliant with oral anticoagulation with either Warfarin, dabigatran, rivoraxaban or apixiban

Exclusion Criteria:

* Inability to follow-up as per protocol
* Prior valvular surgery or valve replacement
* Reversible cause for atrial fibrillation
* Currently on dialysis or renal replacement therapy
* Need for concomitant cardiac surgery
* History of MI or stroke ≤2 months prior to ablation
* Intolerance to oral anticoagulants
* Thrombus in the Left atrial appendage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-12-18 (Estimated)

PRIMARY OUTCOMES:
Number of participants who are free from atrial fibrillation (AF) | 12 months after the procedure

SECONDARY OUTCOMES:
Number of participants who experienced a procedural complication | 2 weeks after the procedure
Number of participants who are at risk of stroke | 12 months after the procedure
Number of participants who were hospitalized for cardiovascular events | 12 months after the procedure
AF burden as assessed by the CCA-SAF | 12 months after the procedure
  AF burden will be assessed using the Canadian Cardiovascular Society - Severity of Atrial Fibrillation Score (CCA-SAF), which provides objective symptoms severity scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Venkataraman, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No